CLINICAL TRIAL: NCT04489147
Title: Effect of Metformin on Non PCO Women Undergoing IVF/ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amira S Dieb, Assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #FWA00015574
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Infertility
Keywords: non PCO
MeSH Terms: conditions — Infertility | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin (Active Comparator): Group A ( involve 200 patients ) will receive metformin 850 mg twice daily along the cycle of ICSI
  Interventions: Drug: Metformin
- No Metformin (No Intervention): Group B ( involve 200 patients) will not receive metformin

INTERVENTIONS:
Drug: Metformin — metformin 850 mg orally twice daily along the cycle of ICSI
  Arms: metformin

SUMMARY:
400 Patients will be randomly assigned into two groups after informed consent from every patient.

They will be classified into 2 groups:

Group A ( involves 200 patients ) will receive metformin 850 mg twice daily along the cycle of Intra-cytoplasmic sperm injection (ICSI) Group B ( involve 200 patients) will not receive metformin. They will undergo a cycle of ICSI. Primary outcome of this trial is to detect occurrence of Ovarian Hyper-stimulation Syndrome (OHSS) , while secondary outcomes include quality & number of retrieved

follicles fertilization rate ,ongoing pregnancy rate & endometrial thickness.

DETAILED DESCRIPTION:
This study is a prospective, single-blinded (to the outcomes assessor), randomized controlled trial conducted at the In Vitro Fertilization ( IVF) centers of the Departments of Obstetrics & Gynecology, Kasr El-Ainy Hospital and Beni-suef hospital in Cairo University and Beni-suef university,respectively, Egypt, to determine the clinical effect of metformin on ICSI outcomes in non PCO patients. Ethical committee approval was obtained. The study will include 400 infertile patients.

Inclusion criteria :

* Patients subjected to IVF/ICSI aged 20-35 years with long agonist protocol
* history of infertility for at least two years (either primary or secondary)
* normal Thyroid stimulating Hormone (TSH) and prolactin

Exclusion criteria :

* Patients who used metformin in the past 3-months before study
* having medical problems such as kidney or liver diseases
* Severe endometriosis.
* hypo-thalamic amenorrhea.
* Severe male factor( patients with testicular biopsy or those with azoo-spermia).
* Associated uterine factor.
* IVF/ ICSI for sex selection. All patients are informed about the study and consent is given by those who accept to participate.

Careful history taking include infertility type, duration , cause, obstetric history, medical and surgical history and demographic distribution is taken. Full physical examination and 2 dimensional (2D) transvaginal sonography (TVS) are done on day 2 to 5 of menses to assess antral follicle count, uterus and adnexa . Body mass index (BMI) and waist/hip ratio (WHR) are calculated, Blood samples are taken for AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2), thyroid stimulating hormone ( TSH), Prolactin and free testosterone.

All 400 participants will be randomized by withdrawing closed envelopes for each patient into group A and group B .

Group A ( involves 200 patients ) will receive metformin 850 mg twice daily along the cycle of ICSI Group B ( involve 200 patients) will not receive metformin.

They will undergo a cycle of ICSI.The agonist protocol is followed.Long protocol steps:

* Start from day 19th - 20th by GnRH agonist ;Triptorelin 0.1mg subcutaneous (Decapeptyl, Ferring). -1st visit : after 2 weeks of start of GnRH agonist or day 2 of cycle, we confirm down regulation by a serum level of E2to be <50 pg/ml, endometrial thickness <5mm, no ovarian cyst by ultrasound. Then we add Gonadotropins as Intramuscular (I.M.) injections of 150-300 I.U. of highly purified Human Menopausal Gonadotropins daily (Merional, 75 I.U. /vial, IBSA). The dose is adjusted according to the age, BMI, AFC, serum levels of anti-mullerian hormone (AMH), follicle stimulating hormone (FSH) and ovarian response.
* 2nd visit : on 6th - 7 th days of Gonadotrophins and then every other day to do folliculometry by TVS and E2 level in serum.
* We do trigger by Human Chorionic Gonadotrophin (HCG)10000 IU I.M.(Pregnyl, Organon) when at least 3 follicles reach 18mm in mean diameter or more and E2 level is less than 2500 pg/ml. Ovum pickup is done 34 hours after HCG injection and embryo transfer using Wallace catheter on day 2 to 3.

  * -Luteal support: Natural Progesterone 400 mg 1x2, Folic acid once daily, Amoxicillin-Clavulanic Acid 1gm 1x2x7 ,Progesterone 100mg I.M. daily for 10 days, Acetylsalicylic Acid once daily
  * -Quantitative ß- HCG in serum after 14 days of embryo transfer. -TVS to detect clinical pregnancy at 6-7 weeks of gestation.

Primary outcome of this trial is to detect occurrence of Ovarian Hyper-stimulation Syndrome (OHSS) , while secondary outcomes include quality & number of retrieved follicles fertilization rate ,ongoing pregnancy rate & endometrial thickness.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to IVF/ICSI aged 20-35 years with long agonist protocol
* history of infertility for at least two years (either primary or secondary)
* normal TSH and prolactin

Exclusion Criteria:

* Patients who used metformin in the past 3-months before study
* having medical problems such as kidney or liver diseases
* Severe endometriosis.
* hypothalamic amenorrhea.
* Severe male factor( patients with testicular biopsy or those with azoospermia).
* Associated uterine factor.
* IVF/ ICSI for sex selection.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Rate of OHSS | 4weeks
  The number of cases of Ovarian Hyperstimulation Syndrome per cycle

SECONDARY OUTCOMES:
The number of Mature retrieved eggs ( M-I) follicles . | 2-4weeks
  The number of mature retrieved eggs (M-I) and each number
fertilization rate | 4weeks
  The number of fertilized eggs after injection with sperms
pregnancy rate | 4 weeks
  number of pregnancies out of all ICSI cycles

CONTACTS AND LOCATIONS:
Overall Officials: Amal Kotb, MD, Study Director — Beni-Suef University
Locations (1):
- Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No